CLINICAL TRIAL: NCT01864798
Title: A Pre-Operative Window Study Evaluating Denosumab, a RANKligand (RANKL) Inhibitor and Its Biological Effects in Young Premenopausal Women Diagnosed With Early Breast Cancer
Brief Title: A Study to Evaluate Denosumab in Young Patients With Primary Breast Cancer
Acronym: D-Beyond
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Jules Bordet Institute (Other)
Collaborators: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-BCTL- 20119167; 2011-006224-21 (EudraCT Number)
Record Dates: First submitted 2013-05-21; First posted 2013-05-30 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Breast Neoplasms
Keywords: Young; Breast Neoplasms; Denosumab; RANKL
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Denosumab (Experimental)
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab
  Other Names: XGEVA

SUMMARY:
This is a prospective, single arm phase IIa trial in which patients with early breast cancer will receive pre-operatively two doses of denosumab 120mg subcutaneously one week apart (maximum 12 days) followed by surgery. Tumor, normal breast tissue and blood samples will be collected at baseline and at surgery. Post-operative treatment will be at the discretion of the investigator.

Primary objective: to determine if a short course of RANKL inhibition with denosumab can induce a decrease in tumor proliferation rates as determined by Ki67 immunohistochemistry (IHC) in newly diagnosed, early stage breast cancer in pre-menopausal women.

Secondary objectives:

* To determine the number of absolute Ki67 responders after a short course of denosumab (defined as <2.7% IHC staining in the post treatment tumor biopsy).
* To determine the effects of a short course of denosumab on serum C-terminal telopeptide levels (CTX).
* To determine the effects of a short course of denosumab on RANK/RANKL gene expression and signaling as assessed by immunohistochemistry (IHC) and RNA sequencing in the tumor.
* To determine the effect of a short course of denosumab on tumor apoptosis rates using IHC
* To determine the effect of a short course of denosumab on modulating the immature mammary epithelial cell populations in the tumor.
* To determine the effect of a short course of denosumab on estrogen signaling pathways in the tumor.
* To determine the effect of a short course of denosumab on various immune
* To determine effect of safety profile of denosumab

ELIGIBILITY:
Inclusion Criteria:

1. Female gender
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Premenopausal status defined as the presence of active menstrual cycle or normal menses during the 6 weeks preceding the start of study treatment. Biochemical evidence of phase of menstrual cycle is required (estradiol, FSH and LH). In women previously exposed to hysterectomy,or were using hormonal intrauterine device at the time of enrolment, premenopausal levels of estradiol, FSH and LH are required to be eligible
5. Non-metastatic operable newly diagnosed primary invasive carcinoma of the breast that is:

   1. Histologically confirmed
   2. Primary tumor size greater than 1.5 cm, measured by any of clinical examination, mammography, ultrasound or magnetic resonance imaging
   3. Any clinical nodal status
   4. Fully operable and not fixed to chest wall.
6. Known HER2 status
7. Known estrogen receptor (ER) status and progesterone receptor status (PgR)
8. Patient has adequate bone marrow and organ function as shown by:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L
   * Hemoglobin (Hgb) ≥ 9.0 g/dL
   * Serum creatinine ≤ 1.5 x ULN
   * Total serum bilirubin ≤ 1.5 x ULN (in patients with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN, with direct bilirubin ≤ 1.5 x ULN)
   * AST and ALT ≤ 1.5 x ULN
   * Random blood sugar (RBS) ≤ 200 mg/dL or ≤ 11.1 mmol/L
   * Glycosylated hemoglobin (HbA1c) ≤ 8 %
9. Albumin-adjusted serum calcium ≥ 8.0 mg/dL (≥ 2.0 mmol/L)
10. Women of childbearing potential must agree to use an active local contraception method for the duration of the study and for at least 7 months after the last dose of study treatment
11. Patients must accept to take calcium and vitamin D supplementation until the completion of the study treatment
12. Signed informed consent form (ICF) for all study procedures according to local regulatory requirements prior to beginning of the study
13. Patients must accept to make available tumor and normal tissue samples for submission to central laboratory at the Jules Bordet Institute, Brussels, Belgium, to conduct translational studies as part of this protocol.

Exclusion Criteria:

1. History of any prior (ipsi and/or contralateral) breast cancer
2. Any "clinical" T4 tumor defined by TNM including inflammatory breast cancer
3. History of non-breast malignancies within the 5 years prior to study entry (except carcinoma in situ of the cervix, of the colon, melanoma in situ and basal cell and squamous cell carcinomas of the skin)
4. Prior or planned systemic anti-cancer therapy before definitive surgery
5. Unhealed or planned dental/oral surgery, current or previous osteonecrosis or osteomyelitis of the jaw
6. Pregnant or lactating women or women of childbearing potential without a negative serum or urinary pregnancy test within 7 days prior to starting study treatment; irrespective of the method of contraception used
7. Active Hepatitis-B virus (HBV), Hepatitis-C virus (HCV) or human immunodeficiency virus (HIV) infection
8. Known hypersensitivity to denosumab
9. Bilateral invasive tumors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Geometric mean change in tumor Ki67 expression | Baseline and surgery at Day 10
  Assessed by immunohistochemistry (IHC) from

SECONDARY OUTCOMES:
Absolute Ki67 responders | Baseline and surgery at Day 10
  KI 67 responders will be defined as below 2.7% Ki67 IHC staining in the post treatment tumor biopsy
C-terminal telopeptide (CTX) serum levels | Baseline and surgery at Day 10
RANK/RANKL gene expression and signalling | Baseline and surgery at Day 10
  Assessed by immunohistochemistry (IHC) and RNA sequencing profile in the tumor
gene expression (AURKA, Ki-67,GGI) | Baseline and surgery at Day 10
  Change in tumor proliferation rates using gene expression (single genes and gene modules, i.e. AURKA, Ki-67) and proliferation-related gene modules, i.e. GGI) in the tumor from baseline to prior to surgery
TUNEL and caspase-3 apoptosis markers | Baseline and surgery at Day 10
  Change in tumor apoptosis rates as measured using TUNEL and caspase-3 IHC from baseline to prior to surgery
expression of immature mammary epithelial cell population: MaSCs, luminal progenitors , ALDH1 | Baseline and surgery at Day 10
  Change in expression levels from genes corresponding to immature mammary epithelial cell populations (MaSCs and luminal progenitors developed by Lim et al; Nature 2009), and in IHC expression of ALDH1, a stem cell marker in the tumor
gene expression of the estrogen pathways (i.e. ESR1, PgR, BCL2) and estrogen-related gene expression modules (i.e. ESR module) | Baseline and surgery at Day 10
  Change in expression levels from single genes related to the estrogen pathways (i.e. ESR1, PgR, BCL2 using both gene expression and IHC) and estrogen-related gene expression modules (i.e. ESR module) in the tumor
immune related genes | Baseline and surgery at Day 10
  Change in expression levels from single genes related to immune pathways using both gene expression and IHC, and in immune-related gene expression modules, to explore the hypothesis that RANKL can modulate T regulatory cells in the tumor
Quantity of tumor infiltrating lymphocytes | Baseline and surgery at Day 10
  Change in the quantity of tumor infiltrating lymphocytes as measured by percentage infiltration of surrounding tumor stroma and intra-tumoral on the H&E slide pre and post treatment
Safety and tolerability of a short course of denosumab | Day 1, day 8 and surgery Day 10

OTHER OUTCOMES:
PgR status (positive vs. negative) | Baseline and surgery at Day 10
RANKL status (IHC positive vs. negative) in normal breast tissue | Baseline and surgery at Day 10
RANKL status (IHC positive vs. negative) in infiltrating cells or stroma | Baseline and surgery at Day 10
RANKL status (IHC positive vs. negative) in tumor tissue | Baseline and surgery at Day 10
RANK status (IHC positive vs. negative) in normal tissue | Baseline and surgery at Day 10
RANK status (IHC positive vs. negative) in tumor tissue | Baseline and surgery at Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Martine J Piccart, Prof., Study Chair — Jules Bordet Institute; Christos Sotiriou, MD, Principal Investigator — Jules Bordet Institute; Hatem Azim, MD, Principal Investigator — Jules Bordet Insitute; Sherene Loi, MD,PhD, Principal Investigator — Melbourne Health
Locations (6):
- Royal Melbourne Hospital, Victoria, Australia
- Belgium (5):
  - Institute Jules Bordet, Brussels
  - Hopital Erasme, Brussels
  - UZ Leuven, Leuven
  - CHU Ambroise Paré, Mons
  - CMSE, Namur

REFERENCES:
- [Derived] Gomez-Aleza C, Nguyen B, Yoldi G, Ciscar M, Barranco A, Hernandez-Jimenez E, Maetens M, Salgado R, Zafeiroglou M, Pellegrini P, Venet D, Garaud S, Trinidad EM, Benitez S, Vuylsteke P, Polastro L, Wildiers H, Simon P, Lindeman G, Larsimont D, Van den Eynden G, Velghe C, Rothe F, Willard-Gallo K, Michiels S, Munoz P, Walzer T, Planelles L, Penninger J, Azim HA Jr, Loi S, Piccart M, Sotiriou C, Gonzalez-Suarez E. Inhibition of RANK signaling in breast cancer induces an anti-tumor immune response orchestrated by CD8+ T cells. Nat Commun. 2020 Dec 10;11(1):6335. doi: 10.1038/s41467-020-20138-8. PMID 33303745